CLINICAL TRIAL: NCT01133769
Title: Operative Versus Non-Operative Treatment For Clavicle Fracture in the PolyTrauma Patient With Associated Chest Injury. A Prospective, Randomized Clinical Trial
Brief Title: Operative Versus Non-Operative Treatment of Clavicle Fracture in PolyTrauma
Status: Withdrawn | Type: Observational
Why Stopped: Institutional issues Institution issues
Sponsor: Anna Rockich (Other)
Collaborators: Synthes Inc. (Industry)
Responsible Party: Sponsor-Investigator, Anna Rockich, Director, General Surgery Clinical Research Program, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: SAH 1198
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2012-05

CONDITIONS: Clavicle Fracture; Chest Injury
Keywords: Clavicle fracture; fixation; polytrauma; Clavicle fracture patients with chest injury
MeSH Terms: conditions — Thoracic Injuries; Multiple Trauma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Surgical vs Non surgical: This is an open, prospective, randomized, dual arm, parallel group clinical study of open reduction and internal fixation (ORIF) or intramedullary nail (IMN) versus non operative treatment for clavicle fracture in polytrauma patients with associated chest injury, with or without additional injuries to the head, abdomen, pelvis and extremities.

SUMMARY:
About 90% of chest injuries in America are due to blunt forces, mostly as a result of motor vehicle collisions and falls. Severity varies from minor bruising to severe chest injuries. For several years, clavicle ("collarbone") fractures have been treated without surgery (non-operatively), even when the fracture is out of place (displaced). Over the last few years, however, treatment has changed more towards surgical fixation (operative), because of the sometimes difficult healing in clavicle fractures that are displaced. Several research studies have shown that cases in which the clavicle fracture never heals completely (non-union) are more frequent after nonoperative treatment, compared to operative fixation. In those cases, surgery is still required, only later (secondary surgery). Further, clavicle malunion, in which the fracture heals but is still out of place) has been shown to be high after nonoperative treatment. Recent published research studies have shown better function, higher patient satisfaction, earlier return to activity (use of the arm) and decreased nonunion and malunion following surgery, also called open reduction/internal fixation. Despite recent published research, there is still a lack of agreement on when surgical fixation should be performed for clavicle fractures.

Patients with chest injuries often have clavicle fractures. Chest injuries can restrict patients' ability to breathe, cough, stand, walk and leave the hospital. Although it is unusual that chest injuries can be improved with surgery, patients with clavicle fractures and chest injuries might recover faster if the clavicle fractures were repaired.

Patients are being asked to take part in the study they have sustained a clavicle fracture associated with a chest injury with or without any other injury to the abdomen, or arms or legs. The aim of this study is to determine the difference in the hospital length of stay, intensive care unit length of stay, respiratory rehabilitation (recovery of good respiratory function), functional outcome, ability to become mobile again, complications and risk of dying in trauma patients with chest injury and clavicle fracture treated operatively versus non-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients males and females of any race.
2. Patients between ages 18 and 80
3. Patients who present with a unilateral clavicle fractures which are >2cm displaced, >2cm shortened, significantly comminuted, or are tenting the skin or which are bilateral and with associated chest injury and with or without additional injuries to the abdomen, pelvis or extremities will be approached for the study.

Exclusion Criteria:

1. Severe brain injury (GCS less than or equal to 13)
2. Intubated patients
3. Injury precluding operative fixation within 7 days of admission
4. Open clavicle fracture
5. Spinal cord injuries
6. Age <18 or greater than or equal to 80

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present with a unilateral clavicle fractures which are >2cm displaced, >2cm shortened, significantly comminuted, or are tenting the skin or which are bilateral and with associated chest injury and with or without additional injuries to the abdomen, pelvis or extremities will be approached for the study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Rowland, M.D., Principal Investigator — St. Anthony's Hospitals/Panorama Orthopedics and Spine Center
Locations (1):
- St. Anthony's Hospitals Centura Health, Denver, Colorado, United States